CLINICAL TRIAL: NCT04480684
Title: A Prospective Observational Study Evaluating the Sonographic Appearance of the Anal Sphincter in Women With Perineal Wound Infection Following Vaginal Delivery.
Brief Title: The Effect of Perineal Wound Infection on the Anal Sphincter
Status: Completed | Type: Observational
Sponsor: Croydon Health Services NHS Trust (Other)
Responsible Party: Principal Investigator, Mr Abdul H Sultan, Consultant Obstetrician & Gynaecologist, Croydon Health Services NHS Trust
Other Study IDs: 278466
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Obstetric Trauma; Perineum; Injury; Perineal Infection; Anal Sphincter Injury
Keywords: Obstetric Anal Sphincter Injury; Childbirth related perineal trauma; Perineal wound infection; Endoanal ultrasound; Transperineal ultrasound; 3D Ultrasound; 4D Ultrasound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Three-dimensional Endoanal Ultrasound — Three-dimensional endoanal ultrasound is the gold standard diagnostic tool in the assessment of obstetric anal sphincter injury. The anorectal transducer is inserted directly into the anal canal which allows assessment of the anal sphincter complex.
  Patients will be assessed at weekly intervals with until the wound infection has resolved and the wound has clinically healed.
Diagnostic Test: Transperineal Ultrasound(multiplanar) — If endoanal ultrasound is declined or not tolerated, the anal sphincter will also be assessed using three-/four-dimensional (3D/4D) transperineal ultrasound with the probe placed externally on the area of the fourchette.
  Patients will be assessed at weekly intervals with until the wound infection has resolved and the wound has clinically healed.
Diagnostic Test: The MolecuLight i:X: Bacterial autofluorescence camera — The bacterial load of the perineal wound will be measured every week using the MolecuLight i:X. This is a system, which uses fluorescent illumination to capture and document the presence of bacteria.
  Patients will be assessed at weekly intervals with until the wound infection has resolved and the wound has clinically healed.
  These findings will be supported by microbiological analysis of the wound fluid with swab culture and sensitivity.
Device: Silhouette® 3D camera: Three-dimensional wound measuring camera — For wound that have superficially dehisced, the wound surface area, depth, volume and healing progress will be precisely measured using the Silhouette® 3D camera. This is a system that uses 3D laser technology to track wound healing progression.

SUMMARY:
Perineal injury following childbirth can result in complications such as wound infection. The perineum has closely related anatomical structures including the external genital organs and the anal triangle which contains the anal sphincter muscles. Therefore as wound infection can extend and as muscles of the perineum sit in such close proximity to each other, the anal sphincter muscles could potentially be affected. This could also potentially include cases of perineal injury where the anal sphincter was not injured.

However ultrasound has never been used to investigate this. Endoanal ultrasound is the gold standard diagnostic tool in the assessment of obstetric anal sphincter injury. The anal sphincter can also be visualised using multiplanar transperineal ultrasound(three/four-dimensional. Therefore both modalities could be used. However, it has been shown that transperineal ultrasound has a high positive predictive value and therefore is able to correctly identify an intact anal sphincter, but low positive predictive value; meaning poor detection of sphincter defects. Therefore, although it cannot completely substitute endoanal ultrasound (the gold standard in investigating obstetric anal sphincter injuries), it provides and adjunct/alternative for women who cannot tolerate endoanal ultrasound.

The investigators plan to perform an observational study to evaluate to the natural history of perineal wound infections. Patients will be assessed weekly with endoanal ultrasound and/or transperineal ultrasound until the wound infection has resolved and the wound has clinically healed.

If a bacterial wound swab has not been taken prior to recruitment or wound swab results are not available, one will be taken to detect the causative organisms. Appropriate antibiotics will then be given to cover the detected organism.

Bacterial burden and will also be measured weekly using the MolecuLight i:X; a bacterial autofluorescence camera which captures the presence and load of bacteria.

In wounds that have superficially dehisced; exact wound measurements including wound surface area, depth, volume and healing progress will be precisely measured using the Silhouette® 3D camera

ELIGIBILITY:
Inclusion Criteria:

* Women with childbirth related perineal injury and wound infection
* Women over 18 years of age
* Ability to understand and read the patient information sheet (in English)
* Ability to give informed consent

Exclusion Criteria:

* Vulnerable Adult
* Fetal or neonatal death or poor neonatal outcome
* Women who are in an immunosuppressive state (e.g human immunodeficiency virus or pharmacologically induced immunodeficiencies by chemotherapy or steroids)
* Inability to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have been referred to the Croydon University Hospital dedicated perineal clinic with perineal wound infection will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Change in sphincter defect 3-point radial angle | Baseline until wound infection resolved and wound healed, or up to 16 weeks
  Endoanal ultrasound and/or transperineal ultrasound will be performed to assess involvement of the anal sphincter.
  Anal sphincter defects will measured on both modalities with a 3-point angle, with the angle vertex in the middle of the anal canal. The 3D volume will be assessed at the deep, superficial, and subcutaneous levels for defects. A change in radial angle size will be measured.
  On transperineal ultrasound the extent of the defect will be measured circumferentially using a 3-point radial angle(0 degrees being no defect). A change in radial angle size will be measured.
Change in sphincter defect Stark Score | Baseline until wound infection resolved and wound healed, or up to 16 weeks
  On endoanal ultrasound, anal sphincter defects will also be scored using a validated Starck score which accounts for depth, length and size of the defect for both internal and external anal sphincter, with a range from 0 being no defect to 16 being maximal defect. Therefore, a change in this score will be measured.

SECONDARY OUTCOMES:
Change in bacterial fluorescence patterns | Baseline until wound infection resolved and wound healed, or up to 16 weeks
  The bacterial load of the perineal wound will be measured every week using the MolecuLight i:X. This is a system, which uses fluorescent illumination to capture and document the presence of bacteria.
Change in wound dimensions | Baseline until wound infection resolved and wound healed, or up to 16 weeks
  Change in total wound size using the Silhouette® 3D camera.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul H Sultan, MB.ChB, MD, FRCOG, Principal Investigator — Croydon Health Services NHS Trust
Locations (1):
- Croydon University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCandlish R, Bowler U, van Asten H, Berridge G, Winter C, Sames L, Garcia J, Renfrew M, Elbourne D. A randomised controlled trial of care of the perineum during second stage of normal labour. Br J Obstet Gynaecol. 1998 Dec;105(12):1262-72. doi: 10.1111/j.1471-0528.1998.tb10004.x. PMID 9883917
- [Background] Royal College of Obstetricians and Gynaecologists (RCOG). Methods and Materials used in Perineal repair, Guideline No 23. London: Royal College of Obstetricians and Gynaecologists Press; 2004.
- [Background] Thakar R, Fenner DE. Anatomy of the Perineum and the Anal Sphincter. In: Sultan AH, Thakar R, Fenner DE, editors. Perineal and Anal Sphincter Trauma: Diagnosis and Clinical Management [Internet]. London: Springer London; 2007. p. 1-12. Available from: https://doi.org/10.1007/978-1-84628-503-5_1
- [Background] Sultan AH. Obstetric Perineal Injury and Anal Incontinence. AVMA Medical & Legal Journal. 1999 Nov;5(6):193-6
- [Background] Webb S, Sherburn M, Ismail KM. Managing perineal trauma after childbirth. BMJ. 2014 Nov 25;349:g6829. doi: 10.1136/bmj.g6829. No abstract available. PMID 25425212
- [Background] Arendsen L, Thakar R, Sultan A. Can perineal wound infection following vagina delivery be reduced? A double blind randomised controlled trial using copper impregnated maternity sanitary towels. European Journal of Obstetrics & Gynecology and Reproductive Biology. 2019 Mar;234:e180.
- [Background] Taithongchai A, van Gruting IMA, Volloyhaug I, Arendsen LP, Sultan AH, Thakar R. Comparing the diagnostic accuracy of 3 ultrasound modalities for diagnosing obstetric anal sphincter injuries. Am J Obstet Gynecol. 2019 Aug;221(2):134.e1-134.e9. doi: 10.1016/j.ajog.2019.04.009. Epub 2019 Apr 11. PMID 30981717
- [Background] European Centre for Disease Prevention and Control. Stockholm. Surgical site infections. In:ECDC. Annual epidemiological report for 2017. 2019.
- [Background] Sultan AH, Kamm MA. Faecal incontinence after childbirth. Br J Obstet Gynaecol. 1997 Sep;104(9):979-82. doi: 10.1111/j.1471-0528.1997.tb12052.x. No abstract available. PMID 9307520
- [Background] National Healthcare Safety Network, Centers for Disease Control and Prevention. Surgical site infection (SSI) event. [Internet]. 2017. Available from: http://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf.
- [Background] Eisenberg VH, Valsky DV, Yagel S. Transperineal ultrasound assessment of the anal sphincter after obstetric anal sphincter injury (OASI). Ultrasound Obstet Gynecol. 2019 Feb;53(2):158-165. doi: 10.1002/uog.19058. No abstract available. PMID 29575180
- [Derived] Okeahialam NA, Thakar R, Sultan AH. Bacterial autofluorescence in infected perineal wounds: A prospective cohort study. Diagn Microbiol Infect Dis. 2023 Jan;105(1):115831. doi: 10.1016/j.diagmicrobio.2022.115831. Epub 2022 Oct 8. PMID 36332560

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT04480684/Prot_SAP_002.pdf
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT04480684/ICF_000.pdf